CLINICAL TRIAL: NCT00256204
Title: A Multi Center, Double Blind, Randomized Start, Placebo-Controlled, Parallel-Group Study to Assess Rasagiline as a Disease Modifying Therapy in Early Parkinson's Disease Subjects
Brief Title: A Randomized Placebo Controlled Study to Show That Rasagiline May Slow Disease Progression for Parkinson's Disease
Acronym: ADAGIO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TVP-1012/500 (ADAGIO)
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Results first posted 2011-06-21 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's; Rasagiline Mesylate
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1mg rasagiline (Experimental): 1mg early start active treatment arm (72 weeks active)followed by 1mg 36 week delayed start active treatment arm (36 weeks placebo followed by 36 weeks active)
  Interventions: Drug: Rasagiline Mesylate
- 2mg rasagiline (Experimental): 2mg early start active treatment arm (72 weeks active)followed by 2mg 36 week delayed start active treatment arm (36 weeks placebo followed by 36 weeks active)
  Interventions: Drug: Rasagiline Mesylate
- Placebo (Placebo Comparator): Each arm is followed by 36 weeks of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rasagiline Mesylate — tablet, 1mg once daily
  Arms: 1mg rasagiline
Drug: Rasagiline Mesylate — tablet, 2mg once daily
  Arms: 2mg rasagiline
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A 2 phase study to evaluate disease progression in Parkinson's disease patients taking rasagiline

ELIGIBILITY:
Inclusion Criteria:

* Men and women with idiopathic PD whose diagnosis is confirmed at screening, with at least two cardinal signs without any other known or suspected cause of parkinsonism. If tremor is not present, subjects must have unilateral onset and persistent asymmetry.
* Subjects with a diagnosis of early idiopathic PD of less than 1½ years duration from time of documented diagnosis.
* Subjects whose clinical condition at the time of enrollment does not require anti-PD treatment and will not require for the next 9 months.
* Willing and able to give informed consent.

Exclusion Criteria:

* Subjects younger than 30 or older than 80 years.
* Subjects with loss of postural reflexes.
* Subjects with UPDRS Tremor score of 3 or greater in any limb.
* Subjects with Hoehn &Yahr Stage III or greater at screening.
* Subjects with freezing while walking.
* Subjects with any of the following features that tend to exclude PD as the cause of Parkinsonism:
* History of repeated strokes with stepwise progression of Parkinsonian features
* History of repeated head injury or history of definite encephalitis
* Sustained remission
* Supranuclear gaze palsy
* Cerebellar signs
* Early severe autonomic involvement
* Babinski's sign
* Presence of a cerebral tumour or communicating hydrocephalus
* MPTP exposure
* Oculogyric crises
* Subjects who have had previous use of rasagiline or selegiline
* Subjects having used other anti-PD medication basis at any time prior to baseline
* Subjects having used other anti-PD medication (including anticholinergics) for less than 3 weeks during the 3 month period prior to baseline. (not including a single L-Dopa dose as part of L-Dopa test)
* Subjects having used any other anti-PD medication (including anticholinergics) for less than 3 weeks prior to the 3 month period preceding baseline whose anti-PD medication is intentionally ceased in order for the subject to enter the study.
* Subjects who have a clinically significant or unstable medical or surgical condition that may preclude safe and complete participation
* Hypertensive subjects whose BP is not well controlled according to the medical record or as observed during the week of home BP recording prior to baseline
* Subjects diagnosed with melanoma based on the screening dermatologic examination, or with a history of melanoma. Subjects with suspicious lesions at baseline who do not undergo biopsy
* Subjects with significant cognitive impairment as defined by MMSE score < 26
* Subjects with clinically significant psychiatric illness, including major depression [Beck Depression Inventory (short form) ≥15
* Subjects with a history of alcohol or substance abuse within the past 2 years
* Subjects who have taken any experimental medications within 60 days prior to baseline
* Subjects who have used coenzyme Q10 (in daily doses > 300 mg) within 120 days prior to baseline
* Subjects who have used sympathomimetics (including over-the-counter remedies - nasal or oral), dextromethorphan, pethidine or St. John's Wort within the 7 days prior to baseline
* Subjects who have used antidepressants within 42 days prior to baseline
* Subjects who have used ciprofloxacin, a potent CYP 1A2 inhibitor within 7 days prior to baseline
* Subjects who have used MAO inhibitors including reserpine or methyldopa within the three months prior to baseline, or treatment with an anti-emetic or antipsychotic medication with central dopamine antagonist activity within the six months prior to baseline
* Women who are not postmenopausal, surgically sterilized, or using adequate birth control [oral birth control pills, IUD, or a long acting injectable form of contraception; barrier methods alone (i.e., condom) are not sufficient]. Women of childbearing potential without a negative pregnancy test at screening. Nursing women

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1174 (Actual)
Dates: Start 2005-11; Primary Completion 2008-04 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoni Weiss, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.

REFERENCES:
- [Derived] Masellis M, Collinson S, Freeman N, Tampakeras M, Levy J, Tchelet A, Eyal E, Berkovich E, Eliaz RE, Abler V, Grossman I, Fitzer-Attas C, Tiwari A, Hayden MR, Kennedy JL, Lang AE, Knight J; ADAGIO investigators. Dopamine D2 receptor gene variants and response to rasagiline in early Parkinson's disease: a pharmacogenetic study. Brain. 2016 Jul;139(Pt 7):2050-62. doi: 10.1093/brain/aww109. Epub 2016 May 13. PMID 27190009
- [Derived] Smith KM, Eyal E, Weintraub D; ADAGIO Investigators. Combined rasagiline and antidepressant use in Parkinson disease in the ADAGIO study: effects on nonmotor symptoms and tolerability. JAMA Neurol. 2015 Jan;72(1):88-95. doi: 10.1001/jamaneurol.2014.2472. PMID 25420207
- [Derived] Rascol O, Fitzer-Attas CJ, Hauser R, Jankovic J, Lang A, Langston JW, Melamed E, Poewe W, Stocchi F, Tolosa E, Eyal E, Weiss YM, Olanow CW. A double-blind, delayed-start trial of rasagiline in Parkinson's disease (the ADAGIO study): prespecified and post-hoc analyses of the need for additional therapies, changes in UPDRS scores, and non-motor outcomes. Lancet Neurol. 2011 May;10(5):415-23. doi: 10.1016/S1474-4422(11)70073-4. Epub 2011 Apr 7. PMID 21482191
- [Derived] Olanow CW, Rascol O, Hauser R, Feigin PD, Jankovic J, Lang A, Langston W, Melamed E, Poewe W, Stocchi F, Tolosa E; ADAGIO Study Investigators. A double-blind, delayed-start trial of rasagiline in Parkinson's disease. N Engl J Med. 2009 Sep 24;361(13):1268-78. doi: 10.1056/NEJMoa0809335. PMID 19776408
- See also: Unified Parkinson's Disease Rating Scale — http://en.wikipedia.org/wiki/Unified_Parkinson's_Disease_Rating_Scale

RESULTS

PARTICIPANT FLOW:
Groups:
- 1mg Delayed Start: 1mg Rasagiline tablet QD 36 week delayed start active treatment arms (36 weeks placebo followed by 36 weeks Rasagiline)
- 1mg Early Start: 1mg Rasagiline tablet QD early start active treatment arm (72 weeks active)
- 2mg Delayed Start: 2mg Rasagiline tablet QD 36 week delayed start active treatment arms (36 weeks placebo followed by 36 weeks Rasagiline)
- 2mg Early Start: 2mg Rasagiline tablet QD early start active treatment arm (72 weeks active)
Period: Overall Study
Arm/Group | 1mg Delayed Start | 1mg Early Start | 2mg Delayed Start | 2mg Early Start
Started | 298 | 288 | 295 | 293
Completed | 231 | 238 | 241 | 244
Not Completed | 67 | 50 | 54 | 49
Not completed — Adverse Event | 10 | 14 | 16 | 14
Not completed — Death | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 2
Not completed — Protocol Violation | 1 | 0 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 17 | 6 | 7 | 5
Not completed — Need for additional prohibited treatment | 38 | 28 | 27 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1mg Delayed Start | 1mg Early Start | 2mg Early Start | 2mg Delayed Start | Total
Number analyzed (Participants) | 298 | 288 | 293 | 295 | 1174
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 175 | 163 | 169 | 173 | 680
  >=65 years | 123 | 125 | 124 | 122 | 494
Age Continuous [Mean (Standard Deviation); unit: years] | 61.9 (9.6) | 62.4 (9.7) | 62.3 (9.6) | 62.4 (9.7) | 62.2 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 113 | 118 | 113 | 457
  Male | 185 | 175 | 175 | 182 | 717
Region of Enrollment [Number; unit: participants]
  United States | 102 | 91 | 94 | 98 | 385
  Portugal | 4 | 4 | 4 | 4 | 16
  Spain | 12 | 12 | 12 | 12 | 48
  Austria | 2 | 2 | 2 | 2 | 8
  Israel | 22 | 23 | 21 | 21 | 87
  United Kingdom | 7 | 7 | 9 | 8 | 31
  Italy | 24 | 25 | 28 | 25 | 102
  France | 11 | 11 | 12 | 14 | 48
  Hungary | 8 | 8 | 6 | 7 | 29
  Canada | 28 | 27 | 29 | 25 | 109
  Argentina | 17 | 17 | 16 | 18 | 68
  Romania | 25 | 24 | 25 | 24 | 98
  Germany | 27 | 28 | 26 | 28 | 109
  Netherlands | 9 | 9 | 9 | 9 | 36

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Unified Parkinson's Disease Rating Scale (UPDRS) Score From Baseline
Description: The primary efficacy endpoint was defined as the change in Total UPDRS from Baseline. Subjects were assessed according to the United Parkinson's Disease Rating Scale (UPDRS,(version 3;) Parts I and II are historical data and are designed to rate mentation, behavior and mood; Part III is done as a motor examination at the time of a visit. The UPDRS measures patient status on a scale 0, which is normal or none, to 4, which is severe or the worst scenario.
Time Frame: 12w, 24w, 36w, 42w, 48w, 54w, 60w, 66w, 72w
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | 1mg Delayed Start | 1mg Early Start | 2mg Early Start | 2mg Delayed Start
Number analyzed (Participants) | 298 | 288 | 293 | 295
Scores on a scale
  Week 12 | 0.9 (4.9) | -1.2 (5.6) | -0.7 (4.8) | 0.7 (5.6)
  Week 24 | 3.0 (6.5) | -1.1 (5.6) | -0.5 (5.6) | 2.2 (6.5)
  Week 36 | 3.7 (7.2) | 0.6 (5.9) | 0.8 (6.5) | 3.0 (6.9)
  Week 42 | 2.4 (7.4) | 0.2 (6.7) | 0.4 (7.2) | 1.7 (6.6)
  Week 48 | 1.9 (6.9) | 0.7 (7.0) | 0.5 (7.1) | 1.4 (6.8)
  Week 54 | 1.9 (7.3) | 0.7 (7.1) | 0.8 (7.2) | 1.1 (7.0)
  Week 60 | 1.9 (7.5) | 1.1 (7.3) | 1.2 (7.9) | 1.6 (7.4)
  Week 66 | 2.5 (8.1) | 1.5 (7.7) | 1.5 (8.0) | 2.0 (8.2)
  Week 72 | 3.3 (8.9) | 1.9 (8.1) | 2.2 (8.1) | 2.3 (7.8)
Statistical Analysis 1: Comparison: 1mg Delayed Start vs 1mg Early Start vs 2mg Delayed Start; Hypothesis #1: Slopes Superiority of 1mg Rasagiline over Placebo in the PC Phase Where slope is the model estimate of the change from baseline in total UPDRS per week. In this analysis, all available post-baseline observations in the PC Phase of the trial are analyzed (ITT efficacy data analysis set, weeks 12, 24 and 36). The placebo groups for rasagiline 1mg (delayed-start) and 2mg (delayed-start)are combined to one placebo group; Test type: Superiority or Other; p = 0.0133, Repeated Measures Mixed Linear Model
Statistical Analysis 2: Comparison: 1mg Delayed Start vs 2mg Early Start vs 2mg Delayed Start; Hypothesis #1: Slopes Superiority of 2mg Rasagiline over Placebo in the PC Phase Where slope is the model estimate of the change from baseline in total UPDRS per week. In this analysis, all available post-baseline observations in the PC Phase of the trial are analyzed (ITT efficacy data analysis set, weeks 12, 24 and 36). The placebo groups for rasagiline 1mg (delayed-start)and 2mg (delayed-start) are combined to one placebo group; Test type: Superiority or Other; p = 0.0001, Repeated Measures Mixed Linear Model
Statistical Analysis 3: Comparison: 1mg Delayed Start vs 1mg Early Start; Hypothesis #2: Superiority of Early over Delayed Start at Week 72 In this analysis, observations of subjects entering the active phase with at least 24 weeks of treatment during the PC Phase and at least one available Total UPDRS measurement during the active-treatment phase from weeks 48, 54, 60, 66 or 72, are analyzed (ACTE data analysis set); Test type: Superiority or Other; p = 0.0250, Repeated Measures — The analysis was performed on separate datasets and not on the combined dataset as was pre-specified to account for unexpected interactions of dose level by baseline UPDRS and of dose level by center
Statistical Analysis 4: Comparison: 2mg Early Start vs 2mg Delayed Start; Hypothesis #2:Superiority of Early over Delayed Start at Week 72 In this analysis, observations of subjects entering the active phase with at least 24 weeks of treatment during the PC Phase and at least one available Total UPDRS measurement during the active-treatment phase from weeks 48, 54, 60, 66 or 72, are analyzed (ACTE data analysis set.); Test type: Superiority or Other; p = 0.6028, Repeated Measures — The analysis was performed on separate datasets and not on the combined dataset as was pre-specified to account for unexpected interactions of dose level by baseline UPDRS and of dose level by center
Statistical Analysis 5: Comparison: 1mg Delayed Start vs 1mg Early Start; Hypothesis #3: Slopes Non-Inferiority of Early Start over Delayed Start in the Active Phase. Where slope is the model estimate of the change from baseline in total UPDRS per week. In this analysis, observations of all subjects entering the active phase with at least 24 weeks of treatment during the PC Phase and at least one available Total UPDRS measurement during the active treatment phase from weeks 48, 54, 60, 66 or 72, are analyzed (ACTE data analysis set); Test type: Non-Inferiority or Equivalence — Non-Inf Test for difference in slopes between treatment groups. One sided 95% CI calculated for difference between slopes of the 1mg early-start group and the 1mg delayed-start group. The inferiority null hypothesis of the early-start group slope over delayed-start group slope is rejected, if the upper limit of one sided 95% CI for difference in slopes does not cross non-inferiority margin of 0.15 UPDRS points per week; Slope = 0.000, 90% CI [-0.036 to 0.036]
Statistical Analysis 6: Comparison: 2mg Early Start vs 2mg Delayed Start; [analysis description as in outcome 1, analysis 5]; Test type: Non-Inferiority or Equivalence — Non-Inf Test for difference in slopes between treatment groups. One sided 95% CI calculated for difference between slopes of the 2mg early-start group and the 2mg delayed-start group. The inferiority null hypothesis of the early-start group slope over delayed-start group slope is rejected, if the upper limit of one sided 95% CI for difference in slopes does not cross non-inferiority margin of 0.15 UPDRS points per week; Slope = 0.029, 90% CI [-0.005 to 0.062]

2. Secondary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS) Score From Baseline to Last Observed Value in the Placebo Phase
Description: Subjects were assessed according to the United Parkinson's Disease Rating Scale UPDRS,(version 3;) Parts I and II are historical data and are designed to rate mentation, behavior and mood; Part III is done as a motor examination at the time of a visit. The UPDRS measures patient status on a scale 0, which is normal or none, to 4, which is severe or the worst scenario.
Time Frame: 36 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- 1mg Delayed Start: + 2 mg Delayed Start: 36 week combined placebo group.
- 1mg Early Start: 1mg early start active treatment arm (72 weeks active)
- 2mg Early Start: 2mg early start active treatment arm (72 weeks active)
- 2mg Delayed Start: +1mg Delayed Start: see 1st column
Arm/Group | 1mg Delayed Start | 1mg Early Start | 2mg Early Start | 2mg Delayed Start
Number analyzed (Participants) | 588 | 286 | 290 | 0
Scores on a scale | 3.9 (7.2) | 1.0 (6.0) | 0.8 (6.5) |
Statistical Analysis 1: Comparison: 1mg Delayed Start vs 1mg Early Start vs 2mg Delayed Start; The adjusted means of the changes in Total UPDRS from baseline to LOV in the placebo-controlled phase, observed in the 1 mg and 2 mg rasagiline early-start groups are compared (two contrasts) to the combined placebo group (1 mg and 2 mg rasagiline delayed-start groups), by applying an Analysis of Covariance model. The model includes treatment group, center and baseline Total UPDRS as covariates. For this analysis, both delayed start arms are pooled as a 'placebo arm'; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -3.005, 95% CI [-3.857 to -2.153]
Statistical Analysis 2: Comparison: 1mg Delayed Start vs 2mg Early Start vs 2mg Delayed Start; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -3.154, 95% CI [-4.004 to -2.305]

ADVERSE EVENTS:
Time Frame: 2 years, 6 months
Description: Each Delayed Start arm was preceded by 36 weeks placebo followed by 36 weeks Rasagiline either 1mg or 2mg; therefore, the placebo groups were combined into one group for the placebo analysis.
Groups:
- Placebo Combined Group: 1mg & 2mg combined placebo group includes those patients in 1mg Delayed start and the 2mg Delayed start arms who received placebo for the first 36 weeks.
- 1mg Active Treatment: 1mg Active & 1mg Delayed. This group includes those patients who received 1mg Rasagiline in both the early start active treatment arm (72 weeks active)and those patients who transitioned to active treatment in the 1mg Delayed start treatment arm (36 weeks active treatment)
- 2mg Active Treatment: 2mg Active & 2mg Delayed. This group includes those patients who received 2mg Rasagiline in both the early start active treatment arm (72 weeks active)and those patients who transitioned to active treatment in the 2mg Delayed start treatment arm (36 weeks active treatment)
Arm/Group | Placebo Combined Group | 1mg Active Treatment | 2mg Active Treatment
Serious Adverse Events (participants affected / at risk) | 22/593 | 37/288 | 44/293
Other Adverse Events (participants affected / at risk) | 82/593 | 40/288 | 34/293
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Combined Group (N=593) | 1mg Active Treatment (N=288) | 2mg Active Treatment (N=293)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina Pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Atrial Fibrilation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vitreous Haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid Ptosis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Parasthesia Oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Chest Discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 4 (4) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 1 (2) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle Hemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3)
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Thyroid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Endometrial Cancer Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung Adenocarcinoma Metastic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Benign Laryngeal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Rectal cancer Metastic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid Haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lacunar Infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Akinesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Parkinson's Disease (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Major Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Alcohol Abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Renal Colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Laryngeal Leukoplakia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia Facial (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Coronary Artery Bypass (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Cardioversion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Open reduction of fracture (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Incisional Hernia Repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Inguinal Hernia Repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Knee Operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Colon Polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial Ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Retinal Vein Occlusion (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Heus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rectal Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peridiverticular Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Arteriogram Coronary Abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ovarian Epithelial Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostrate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Loss of Consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neurosis (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hallucination, Visual (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Colpocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Infarction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Arterial Stent Insertion (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Coronary Angioplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Bone operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Hip Arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1)
Hip Surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Knee Arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2)
Cataract Operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Transurethral Prostatectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Aortic Aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Aortic Aneurysm Rupture (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Combined Group (N=593) | 1mg Active Treatment (N=288) | 2mg Active Treatment (N=293)
Back Pain (Musculoskeletal and connective tissue disorders) | 32 (34) | 14 (14) | 15 (15)
Headache (Nervous system disorders) | 37 (39) | 14 (15) | 15 (15)
Fatigue (General disorders) | 17 (18) | 17 (18) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should the Oversight Committee wish to publish the results of this study, the Oversight Committee agrees to provide Teva with a manuscript for review 60 days prior to submission for publication. Teva retains the right to delete from the manuscript confidential information and to object to suggested publication and/or its timing (at the sole discretion of Teva).